CLINICAL TRIAL: NCT02755025
Title: Evaluation of Clinical Score Usefulness and Feasibility of Integration Into Electronic Health Record Interfaces
Brief Title: Clinical Score Usefulness and EHR Integration
Acronym: ScoreInt
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher Aakre, Senior Associate Consultant, Mayo Clinic
Other Study IDs: 15-009228
Record Dates: First submitted 2016-03-15; First posted 2016-04-28 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Sepsis
Keywords: Sepsis; SOFA score; Automated calculation
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prospective cohort: This group will include ICU patients for the two month period after the automated SOFA score has been activated within the electronic patient care dashboard.
  Interventions: Other: Automated SOFA scoring calculator

INTERVENTIONS:
Other: Automated SOFA scoring calculator — Automated SOFA scoring will be activated within an existing electronic patient care dashboard for ICU patients.

SUMMARY:
The SOFA score is a severity of illness and prognostic score used in the ICU. It has also recently been adopted as part of the definition of sepsis. This study will prospectively evaluate the usability of automated SOFA scoring for ICU patients within an electronic patient monitoring dashboard. It will also assess for changes in physician ordering (volume and types of orders) after automatic scoring is implemented.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the medical intensive care unit within 2 months of automated SOFA scoring module activation.

Exclusion Criteria:

* Refusal to allow medical records to be used for clinical research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the medical intensive care unit during the 2 month time period after the automated SOFA scoring module is activated within the electronic dashboard.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
SOFA related laboratory order volume | 2 months
  The total number of SOFA related laboratory orders on all patients in the ICU during the intervention period

SECONDARY OUTCOMES:
Module usability | 2 months
  Providers will be surveyed on the usability of the automated scoring module

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Aakre, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No